CLINICAL TRIAL: NCT01925313
Title: A Randomized, Open Label, Three-Treatment, Three-Period, Six-Sequence Crossover Study To Compare Safety and Pharmacokinetic Properties of CJ-30044 and Bepotastine Besilate and To Investigate Food-effect on Pharmacokinetics of CJ-30044 in Healthy Adult Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CJ_BEP_101
Record Dates: First submitted 2013-08-15; First posted 2013-08-19 (Estimated); Last update posted 2013-08-19 (Estimated); Status verified 2012-12

CONDITIONS: Healthy
Keywords: Safety; Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CJ-30044 (Experimental)
  Interventions: Drug: CJ-30044
- TALION TAB. 10mg (Active Comparator)
  Interventions: Drug: TALION TAB. 10mg

INTERVENTIONS:
Drug: CJ-30044 — 20.51mg a day,PO,QD
  Arms: CJ-30044
Drug: TALION TAB. 10mg — 10mg a day,PO,BID
  Arms: TALION TAB. 10mg

SUMMARY:
Study objectives

* To compare the safety and pharmacokinetic properties of CJ-30044 and bepotastine besylate after a single oral administration in healthy male volunteers.
* To evaluate the food-effect on pharmacokinetics of CJ-30044 after a single oral administration in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Male volunteers in the age between 20 and 45 years old

   * BMI(Body Mass Index) in the range of 18.5 to 25kg/m2
2. Subject with no history of any significant chronic disease
3. Judged to be in good health on the basis of their vital sign, ECG, physical exam and routine laboratory data for this trial by investigators
4. Willing to adhere to protocol requirements and sign a informed consent form

Exclusion Criteria:

1. History of clinically significant allergies, including Bepotastine.
2. History of clinically significant hepatic, renal, neurology, psychiatric, pulmonary, endocrine, hematologic, cardiovascular disease
3. History of surgery except or gastrointestinal disease which might significantly change absorption of medicines
4. Subjects considered as unsuitable health on the basis of their vital sign, ECG, physical exam and routine laboratory data for this trial by investigators.
5. Clinical laboratory test values are outside the accepted normal range

   * AST or ALT >1.25 times to normal range
   * Total bilirubin >1.5 times to normal range
6. Estimated GFR(Glomerular Filtration Rate) < 80 mL/min/1.73m2
7. Clinically significant vital sign

   * SBP(Systolic Blood Pressure) ≤ 90 mmHg or SBP ≥ 150 mmHg
   * DBP(Diastolic Blood Pressure) ≤ 50 mmHg or DBP ≥ 100 mmHg
8. History of drug abuse or positive urine screen for drugs
9. History of caffeine, alcohol, smoking abuse

   * caffeine > 5 cups/day
   * alcohol > 210g/week
   * smoking > 10 cigarettes/day
10. Special diet known to interfere with the absorption, distribution, metabolism or excretion of drugs (especially, consumption of grapefruit juice) within 7 days prior to drug administration
11. Use of prescription only medicine and oriental medicine within the 14 days before dosing or use of non-prescription medicine within the 7 days before dosing
12. Participated in a previous clinical trial within 60 days prior to dosing
13. Donated blood within 60 days prior to dosing
14. Subjects considered as unsuitable based on medical judgement by investigators

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-12; Primary Completion 2013-02 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
AUClast and Peak plasma concentration (Cmax) of Bepotastine | Blood sampling up to 36hs post dose.

SECONDARY OUTCOMES:
AUCinf, Tmax, T1/2 of Bepotastine | Blood sampleing up to 36hrs post dose

CONTACTS AND LOCATIONS:
Overall Officials: Min-Su Park, PhD, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei university severance hospital, Seoul, South Korea